CLINICAL TRIAL: NCT01440803
Title: Randomized Controlled Trial of Teriparatide for the Treatment of Idiopathic Osteoporosis in Premenopausal Women
Brief Title: Forteo Trial on Idiopathic Osteoporosis in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Shane (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Elizabeth Shane, Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAF2251; R01FD003902-01 (FDA)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Adult Idiopathic Generalized Osteoporosis
Keywords: osteoporosis; premenopausal; forteo; idiopathic; Idiopathic Osteoporosis in Premenopausal Women
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teriparatide (Forteo) (Active Comparator): Daily injection of Teriparatide for treatment of idiopathic osteoporosis
  Interventions: Drug: Teriparatide
- Placebo saline injection (Placebo Comparator): Daily injection of saline placebo for 6 months, followed by 24 months of teriparatide treatment for idiopathic osteoporosis.
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: Teriparatide — Daily injection of 20 mcg teriparatide for the treatment of idiopathic osteoporosis for 24 months.
  Other Names: Forteo; TPTD
  Arms: Teriparatide (Forteo)
Drug: Saline Placebo — Daily injection of saline placebo for 6 months, followed by teriparatide treatment for 24 months.
  Other Names: Placebo
  Arms: Placebo saline injection

SUMMARY:
Idiopathic osteoporosis (IOP) is defined as osteoporosis that affects young, otherwise completely healthy individuals with no secondary cause of bone loss. In the course of our prior research with premenopausal women with IOP, the investigators have shown that women with IOP have low areal bone mineral density (aBMD) at the spine, hip and forearm compared to normal women. Additionally, using noninvasive high resolution imaging of the central and peripheral skeleton and detailed analyses of transiliac crest bone biopsies, the investigators identified several features of bone quality in premenopausal women with IOP.

There is currently no FDA-approved therapy for IOP in premenopausal women. However, teriparatide (Forteo) has been shown to improve bone mass and microarchitecture in postmenopausal women and is approved for men with primary or idiopathic osteoporosis, as well as men, premenopausal and postmenopausal women with glucocorticoid-induced osteoporosis. Because IOP in premenopausal women is an orphan disease, with an estimated prevalence of about 113,000 in the United States, pharmaceutical companies are unlikely to support development of therapies for this indication. Therefore, the major objective of this protocol is to establish the safety and efficacy of teriparatide in premenopausal women with IOP in a phase 2 clinical trial. All subjects will receive teriparatide as part of the study, but a randomly selected group of patients (10) will receive one year of placebo injections first before starting their two years of treatment. The remainder of subjects (30) will receive active drug only for two years.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Osteoporosis is a skeletal disorder characterized by reduced bone strength that predisposes to an increased risk of fracture. Osteoporosis affects postmenopausal women and elderly men and is very unusual in healthy individuals under age 50. Moreover, more than 90% of young men and premenopausal women with osteoporosis have a secondary cause of bone lose, such as an underlying disorder (e.g., hypogonadism) or a medication exposure (e.g., glucocorticoids, antiepileptic drugs), that either interfered with acquisition of peak bone mass or caused excessive bone loss thereafter. Idiopathic osteoporosis (IOP) is defined as osteoporosis that affects young, otherwise completely healthy individuals with intact gonadal function and no secondary cause of bone loss. First described by Fuller Albright in 1944, IOP is an uncommon condition with an estimated annual incidence of 0.4 cases per 100,0003. IOP predominantly affects Caucasians, who generally present in their mid-30s with one more low trauma fractures.

In the course of a previously conducted NIH-funded study of premenopausal women, the investigators demonstrated that women with IOP have low areal bone mineral density (aBMD) at the spine, hip and forearm compared to normal women. Additionally, using noninvasive high resolution imaging of the central and peripheral skeleton and detailed analyses of transiliac crest bone biopsies, the investigators identified several distinctive and consistent features of bone quality in premenopausal women with IOP: thin cortices, lower trabecular volumetric bone mineral density (vBMD), fewer trabecular plates, fewer and longer trabecular rods, decreased connectivity between rods and plates, lower mineralization density and lower estimated stiffness of cancellous bone. Bone remodeling and biochemical indices of mineral metabolism did not differ between IOP subjects and controls.

Although not every woman with IOP requires pharmacologic intervention, many have sustained multiple low-trauma fractures or have extremely low bone mineral density (BMD). There is currently no FDA-approved therapy for IOP in premenopausal women, therefore a safe and effective therapy is urgently needed. Bisphosphonates are one therapeutic option but the associated gains in BMD are primarily due to reduction in the remodeling space and increased mineralization of bone rather than improvements in microarchitecture, an important consideration as microarchitectural deficits are a consistent feature of IOP in premenopausal women, while remodeling activity is most commonly normal or low. Furthermore, potential teratogenic effects limit the safety of bisphosphonates in premenopausal women.

However, anabolic therapy with human recombinant parathyroid hormone (hPTH) 1-34 (or teriparatide (TPTD)), has been shown to improve bone mass and microarchitecture in postmenopausal women and is approved for men with primary or idiopathic osteoporosis, as well as men, premenopausal and postmenopausal women with glucocorticoid-induced osteoporosis. TPTD, on the other hand, increases bone formation and BMD, while improving microarchitecture and strength. Moreover, TPTD has been shown to increase BMD in men with IOP, in premenopausal women with glucocorticoid-induced osteoporosis (GIOP) and to prevent bone loss in premenopausal women with nafarelin-induced acute estrogen deficiency. Although there have been no studies evaluating TPTD in estrogen-replete premenopausal women with IOP, data from studies of hPTH(1-34) in postmenopausal women on estrogen are relevant to this proposal. These studies found increased aBMD at the LS and of lesser magnitude at the hip, as well as major reductions in vertebral fracture. Also important, BMD remained stable in postmenopausal women on estrogen followed for two years after TPTD discontinuation. Lane et al. reported similar results in postmenopausal women with GIOP on estrogen. These two studies suggest that in estrogen-replete premenopausal women with IOP, increases in bone mass resulting from TPTD will be sustained after the course of therapy is completed.

The major objective of this protocol is a therapeutic one, namely to establish the safety and efficacy of TPTD in premenopausal women with IOP in a phase 2 clinical trial. The investigators hypothesize that anabolic therapy with teriparatide will improve areal and vBMD in premenopausal women with IOP. The investigators also hypothesize that teriparatide will restore abnormal microarchitecture toward normal and improve other aspects of bone quality in premenopausal women with IOP. The primary aim of this research study will be to establish the efficacy and safety of 6 months of teriparatide versus placebo in premenopausal women with IOP. The secondary aim is to determine the extent to which 12 and 24 months of teriparatide improves areal and volumetric BMD, bone microarchitecture and stiffness compared to baseline measures in premenopausal women with IOP. This study will have high impact on clinical practice as it pertains to the management of premenopausal women with IOP.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, aged 20-45, with regular menses and no historical or biochemical secondary cause of osteoporosis.
* Documented adult fractures judged to be low-trauma.
* Must be willing to use effective contraception throughout the period of study drug administration.

Inclusion Criteria - vary slightly based on age category:

* Premenopausal women ages 20-35 years must have at least one major osteoporotic fracture (excluding fractures of fingers, toes and face) and low Bone Mineral Density (BMD).
* Premenopausal women above the age of 35 years should have a history of fracture and/or low BMD.

Exclusion Criteria:

* History of any condition that increases the risk of osteosarcoma
* Early follicular phase serum
* Disorders of mineral metabolism
* Suspicion of osteomalacia
* Vitamin D deficiency
* Pregnancy or lactation within past 12 months
* Prolonged amenorrhea (> 6 months) during reproductive years (except pregnancy or lactation)
* Prior eating disorder
* Malignancy, except cured basal or squamous cell skin carcinoma
* Endocrinopathy: new onset untreated hyperthyroidism, hypothyroidism, Cushing's syndrome, prolactinoma
* Renal insufficiency
* Liver disease
* Intestinal disorders
* History/current glucocorticoids (GCs), anticonvulsants, anticoagulants, methotrexate, depot progesterone, Gonadotrophin-releasing hormone (GnRH) agonists
* Oral glucocorticoid use (subject will not be excluded if used dose equivalent to less than prednisone 5 mg for <3 months).
* Current anticoagulant use or low molecular weight
* Depo Provera use (subjects will not be excluded if used at age>20, >5 years ago)
* Drugs for osteoporosis (raloxifene, bisphosphonates, denosumab, calcitonin, TPTD). Subjects who discontinue these medications will be eligible 3 months after stopping raloxifene or calcitonin, 12 months after stopping alendronate, risedronate, ibandronate, or pamidronate and 18 months after stopping denosumab. Subjects with prior use of zoledronate may be eligible if received only one dose >4 years ago. Total bisphosphonate exposure must be < 1 year. Subjects who have taken TPTD in the past will not be eligible unless used for <3 months, > 2 years ago.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-08-02 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, MD, Principal Investigator — Columbia University; Adi Cohen, MD, Study Director — Columbia University; Emily M Stein, MD, Study Director — Columbia University
Locations (2):
- United States (2):
  - Creighton University, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen A, Shiau S, Nair N, Recker RR, Lappe JM, Dempster DW, Nickolas TL, Zhou H, Agarwal S, Kamanda-Kosseh M, Bucovsky M, Williams JM, McMahon DJ, Stubby J, Shane E. Effect of Teriparatide on Bone Remodeling and Density in Premenopausal Idiopathic Osteoporosis: A Phase II Trial. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3540-56. doi: 10.1210/clinem/dgaa489. PMID 32876328
- [Derived] Cohen A, Kamanda-Kosseh M, Recker RR, Lappe JM, Dempster DW, Zhou H, Cremers S, Bucovsky M, Stubby J, Shane E. Bone Density After Teriparatide Discontinuation in Premenopausal Idiopathic Osteoporosis. J Clin Endocrinol Metab. 2015 Nov;100(11):4208-14. doi: 10.1210/jc.2015-2829. Epub 2015 Sep 10. PMID 26358172
- [Derived] Nishiyama KK, Cohen A, Young P, Wang J, Lappe JM, Guo XE, Dempster DW, Recker RR, Shane E. Teriparatide increases strength of the peripheral skeleton in premenopausal women with idiopathic osteoporosis: a pilot HR-pQCT study. J Clin Endocrinol Metab. 2014 Jul;99(7):2418-25. doi: 10.1210/jc.2014-1041. Epub 2014 Mar 31. PMID 24684466
- [Derived] Cohen A, Stein EM, Recker RR, Lappe JM, Dempster DW, Zhou H, Cremers S, McMahon DJ, Nickolas TL, Muller R, Zwahlen A, Young P, Stubby J, Shane E. Teriparatide for idiopathic osteoporosis in premenopausal women: a pilot study. J Clin Endocrinol Metab. 2013 May;98(5):1971-81. doi: 10.1210/jc.2013-1172. Epub 2013 Mar 29. PMID 23543660
- See also: Columbia University, Dept of Medicine, Division of Endocrinology website — http://columbiamedicine.org/divisions/Endo/index.shtml

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Periods have been added to represent the sequential nature of the study (e.g., "Period 1: Double blind Forteo/Placebo", "Period 2: Double Blind Forteo/Forteo", "Period 3: Open Label Forteo", etc.) per PRS.
Groups:
- Placebo Saline Injection: First 6 months:
  Placebo Saline Injection Group receiving daily injection of saline placebo
  6-12 months: Placebo Saline Injection Group receiving daily injection of Teriparatide for treatment of idiopathic osteoporosis (20 mcg)
  12-24 months: Forteo open label
- Teriparatide (Forteo): First 6 months:
  Teriparatide (Forteo) Group receiving daily injection of Teriparatide for treatment of idiopathic osteoporosis (20 mcg)
  6-12 months: Teriparatide (Forteo) Group receiving daily injection of Teriparatide for treatment of idiopathic osteoporosis (20 mcg)
  12-24 months: Forteo open label
Period: Overall Study
Arm/Group | Placebo Saline Injection | Teriparatide (Forteo)
Started | 13 | 28
Period 1 - Forteo/Placebo | 13 | 28
Period 2 - Forteo/Forteo | 13 | 28
Period 3 - Forteo Open Label | 13 | 27
Completed | 11 | 24
Not Completed | 2 | 4
Not completed — Met study stopping rule | 2 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide (Forteo) | Placebo Saline Injection | Total
Number analyzed (Participants) | 28 | 13 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 13 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 13 | 41
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 12 | 39
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Columbia University | 23 | 9 | 32
  United States: Creighton University | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine Bone Mineral Density (LS-BMD) on Active Medication
Description: Dual Energy X-ray Absorptiometry (DXA) will be used to measuring bone mineral density (BMD).
Time Frame: Baseline and 12 months
Population: One patient in the Teriparatide (Forteo) arm was lost to follow up before the completion of the 12 month visit, therefore could not be analyzed for the primary outcome.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Teriparatide (Forteo) | Placebo Saline Injection
Number analyzed (Participants) | 27 | 13
percentage of change | 10.1 (5.4) | 4.1 (6.5)

ADVERSE EVENTS:
Time Frame: Up to 30 months, with the following time points: 1 week, 1 month, 3 month, 6 month, 9 month, 12 month, 18 month, 24 month, 30 month
Groups:
- Teriparatide (Forteo) (24 Months): Daily injection of 20 mcg teriparatide for the treatment of idiopathic osteoporosis for 24 months.
- Placebo Saline Injection (6 Months): Daily injection of saline placebo for 6 months.
- Placebo Saline Injection (6-24 Months): Daily injection of 20 mcg teriparatide for the treatment of idiopathic osteoporosis for 18 months following placebo.
Arm/Group | Teriparatide (Forteo) (24 Months) | Placebo Saline Injection (6 Months) | Placebo Saline Injection (6-24 Months)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/28 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT01440803/Prot_SAP_000.pdf